CLINICAL TRIAL: NCT00196950
Title: Assess the Safety, Reactogenicity, Immunogenicity & Long-term Persistence of One Intramuscular Dose of GSK Biologicals' MenACWY Conjugate Vaccine vs One Subcutaneous Dose of Mencevax™ ACWY in Healthy Adults Aged 18-25 Yrs
Brief Title: Study to Evaluate Meningococcal Serogroups A,C,W-135,Y Conjugate Vaccine When Given as 1 Dose to Healthy Subjects Aged 18-25 Years
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 134612/003; 102252 (Other: GSK); 102253 (Other: GSK); 102254 (Other: GSK)
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Infections, Meningococcal
MeSH Terms: conditions — Meningococcal Infections | interventions — Meningococcal Vaccines

INTERVENTIONS:
Biological: Meningococcal (vaccine)

SUMMARY:
The purpose of this study is to evaluate the safety, reactogenicity, immunogenicity and persistence up to three years after administration of one dose of the MenACWY conjugate vaccine when given to young adults aged 18-25 years.

DETAILED DESCRIPTION:
Administration of the candidate vaccine or of the active control (Mencevax™ ACWY) will be done in an open manner. The study consists of a vaccination phase during which subjects receive one vaccine dose (GSK's MenACWY conjugate vaccine or Mencevax™ ACWY vaccine) and 3 years of follow-up. There are in total 7 visits to the doctor: before and 2, 7 and 30 days after vaccination (vaccination phase) as well as 12, 24 and 36 months after vaccination (follow-up phase). 7 blood samples are taken: one at each visit.

ELIGIBILITY:
Inclusion criteria:

* Healthy male or female between, and including, 18 and 25 years of age at the time of vaccination.
* Written informed consent obtained.
* Subject with previously completed routine childhood vaccinations to the best of his/her knowledge.
* Female subjects should be of non-childbearing potential, or abstinent, or using an adequate contraception.

Exclusion criteria:

* Previous vaccination against OR history of OR exposure within previous 12 months to, meningococcal serogroup A, C, W-135 or Y disease.
* Administration of a tetanus vaccine within 6 months before study vaccination.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* A family history of congenital or hereditary immunodeficiency.
* History of any neurologic disorders or seizures.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* History of chronic alcohol consumption and/or drug abuse

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2003-09; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
The occurrence of any grade 3 solicited symptoms within 8 days (day 0-7) following vaccination.

SECONDARY OUTCOMES:
Sol (d 0-7, local&general), unsol (d 0-30) symptoms. SAEs. Routine blood & urine examination before, 2&7 d post vacc. % SBA-MenA C W Y responders 1m post vacc. Antibodies to MenA C W Y before, 1, 12, 24&36m post vacc & tetanus before, 1m post vacc

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Gosselies, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Ostergaard L, Lebacq E, Poolman J, Maechler G, Boutriau D. Immunogenicity, reactogenicity and persistence of meningococcal A, C, W-135 and Y-tetanus toxoid candidate conjugate (MenACWY-TT) vaccine formulations in adolescents aged 15-25 years. Vaccine. 2009 Jan 1;27(1):161-8. doi: 10.1016/j.vaccine.2008.08.075. Epub 2008 Oct 1. PMID 18834910
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 134612/003 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 134612/003 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 134612/003 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register. The results of this study 134612/003 are summarised with studies 102252, 102253, and 102254 on the GSK Clinical Study Register.
- Available data/document: Informed Consent Form: 134612/003 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 134612/003 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 134612/003 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register